CLINICAL TRIAL: NCT05092685
Title: Phase I/II Open Label, Multicentre Clinical Trial to Assess Safety and Efficacy of AAVLK03hOTC for Paediatric Patients With Ornithine Transcarbamylase Deficiency.
Brief Title: Halting Ornithine Transcarbamylase Deficiency With Recombinant AAV in ChildrEn
Acronym: HORACE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18/0123
Record Dates: First submitted 2021-09-28; First posted 2021-10-25 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Ornithine Transcarbamylase Deficiency
MeSH Terms: conditions — Ornithine Carbamoyltransferase Deficiency Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AAVLK03hOTC (also known as ssAAV-LK03.hAAT.hcoOTC) (Experimental): Dose escalation in three groups from 6x10^11vg/kg (low dose), 2x10^12vg/kg (intermediate dose) to 6x10^12vg/kg (high dose). Dose expansion in a fourth group with the best acceptable safety:efficacy ratio
  Interventions: Genetic: AAVLK03hOTC

INTERVENTIONS:
Genetic: AAVLK03hOTC — Peripheral intravenous infusion of AAVLK03hOTC.
  Other Names: Also known as ssAAV-LK03.hAAT.hcoOTC

SUMMARY:
Ornithine transcarbamylase deficiency (OTCD) is an inherited metabolic liver disease which means that the body cannot maintain normal levels of ammonia. Ammonia levels can rise (called hyperammonaemic decompensations) which can be life-threatening and may result in impaired neurological development in children. OTCD is a rare genetic disorder characterised by complete or partial lack of the enzyme ornithine transcarbamylase (OTC).

DETAILED DESCRIPTION:
OTC is a key element of the urea cycle, which is how the liver breaks down and removes extra nitrogen from the body. For people with OTCD the extra nitrogen builds up in the form of excess ammonia (hyperammonemia) in the blood.

Ammonia is toxic and people with OTCD suffer 'hyperammonaemic decompensations' when ammonia levels in the blood rise too high. The symptoms of these hyperammonaemic decompensations include vomiting, impaired movement, and progressive lethargy. If left untreated these hyperammonaemic decompensations may result in life-threatening complications or coma. OTCD is managed with drugs that reduce the amount of ammonia in the blood (ammonia-scavenging drugs) and a low protein diet. However, sometimes hyperammonaemic decompensations still occur.

Liver transplants for people with OTCD can be life-saving but there may be a long wait for a suitable liver and neurological damage may occur before a liver transplant is possible.

The HORACE study is testing a new gene therapy (AAVLK03hOTC) which specifically targets the liver so that it can start making OTC. The investigators hope that a single injection of gene therapy for children with OTCD could help the liver work normally and reduce hyperammonaemic decompensations and their associated risks.

This gene-therapy treatment could serve as a 'bridge-to-transplant' where children could grow up in a metabolically stable condition until a liver transplant is possible. This could minimise longer-term neurological damage caused by hyperammonaemic decompensations.

ELIGIBILITY:
Inclusion Criteria:

1. Patient (male or female) aged ≤16 years at time of written informed consent. For the dose escalation phase patients must be aged 6-16, for the dose expansion phase patients must be aged 0-16 (at the time of written informed consent).
2. OTC deficiency confirmed via enzymatic or molecular analysis. This may include identification of pathogenic mutations or liver OTC activity that is <20% of normal activity.
3. Patient has severe disease defined by reduced protein allowance and prescribed at least one ammonia scavenger drug.
4. Patient (if capable of signing) and parents or legal representative have signed a written informed consent form.
5. Females of childbearing potential must have a negative pregnancy test in serum or urine at the screening and Day 0 infusion visits, and use an adequate contraception method from the screening visit until 4 weeks after the first negative plasma sample monitoring vector genomes copies or the week 52 visit, whatever comes first.
6. Sexually active boys must use an adequate contraception method (abstinence or use of condom with spermicide) from at least 14 days prior to the infusion and until 4 weeks after the first negative plasma sample monitoring vector genomes copies or the week 52 visit, whatever comes first.
7. Patient's ammonia level at baseline visit (pre-gene therapy infusion) is <100µmol/L and is within the range of historical ammonia levels obtained when the patient was clinically stable.
8. Patient has been on a stable dose of ammonia scavenger and stable protein allowance for the last 4 weeks at the baseline visit.
9. Patient is willing to commit to an additional 4 years of long-term safety follow-up.

Exclusion criteria:

1. Titres of the neutralising antibodies against AAV-LK03 >1:5 serum dilution.
2. Significant hepatic inflammation as evidenced by the following laboratory abnormalities: alanine aminotransferase or aspartate aminotransferase or bilirubin >2 x upper limit of normal (ULN), alkaline phosphatase >3 x ULN.
3. Evidence of severe unexplained liver disease including but not limited to liver malignancy, liver cirrhosis, or acute liver failure.
4. Evidence of active hepatitis B or C virus (HBV and HCV respectively) documented by hepatitis B surface antigen (HBsAg) or HCV RNA positivity.
5. Positive PCR for human immunodeficiency virus (HIV).
6. Liver transplant including hepatocytes/cells infusion.
7. Current participation in another clinical trial of an investigational medicinal product or medical device, or participation within previous 12 months.
8. Patient has contraindication to immunosuppression.
9. Active infection (bacterial or viral).
10. Pregnant or breastfeeding females.
11. Patients with other serious underlying medical conditions including malignancy and severe (≥ grade 3) functional organ impairment (liver, kidney, respiratory) according to CTCAE v5.0. For neurological symptoms considered as sequelae of previous hyperammonaemic decompensation and which are considered as stable (i.e. not evolving), a grade 3 will be acceptable. Grade 4 and 5 will preclude inclusion.
12. Patients with any other significant condition or disability that, in the investigator opinion, may interfere with the patient's optimal participation in the study.

Ages: 0 Days to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety - adverse events | 12 months post-infusion
  Incidence of adverse events (AEs), treatment-related adverse events and serious adverse events (SAEs) for each dosing group assessed by severity and relationship to study product.

SECONDARY OUTCOMES:
Safety outcomes | Over 12 months post-infusion
  • Change from baseline level of transaminases (AST and ALT).
Safety outcomes | Over 12 months post-infusion
  Change from baseline level of humoral and cellular immune responses the AAV-LK03 capsid.
Safety outcomes | Over 12 months post-infusion
  • Change from baseline level of cellular immune against hOTC.
Safety outcomes | Over 12 months post-infusion
  • Viral shedding: plasma/saliva/urine/stool samples.
Efficacy outcomes | Over 12 months post-infusion
  Clinical parameters
  • Monitoring of number and frequency of hyperammonaemic episodes and hospitalisations
Efficacy outcomes | Over 12 months post-infusion
  Clinical parameters
  • Monitoring of daily protein allowance using the Nutritics food diary app
Efficacy outcomes | Over 12 months post-infusion
  Clinical parameters
  • Monitoring number of ammonia scavenger drugs.
Efficacy outcomes | Over 12 months post-infusion
  Biological parameters
  • Change from baseline levels of glutamine and glutamate.
Efficacy outcomes | Over 12 months post-infusion
  Biological parameters
  • Change from baseline levels of ammonaemia.
Efficacy outcomes | Over 12 months post-infusion
  Biological parameters
  • Change from baseline levels of urine orotic acid.
Efficacy outcomes | Over 12 months post-infusion
  Functional parameters:
  • Change from baseline rate of ureagenesis rate.

OTHER OUTCOMES:
Exploratory outcomes | Over 12 months post-infusion
  • Change from baseline neurocognitive assessment, as measured by the Bayley - III for participants aged 6months to 3 years
Exploratory outcomes | Over 12 months post-infusion
  • Change from baseline neurocognitive assessment as measured WPPSI-IV for participants aged 2 years 6 months to 7 years 7 months
Exploratory outcomes | Over 12 months post-infusion
  • Change from baseline neurocognitive assessment as measured by the WISC-V for participants aged 6 years to 16 years and 11months
Exploratory outcomes | Over 12 months post-infusion
  • Change from baseline behavioural assessment as measured by the Child Behaviour Checklist
Exploratory outcomes | Over 12 months post-infusion
  • Change from baseline in adaptive functioning, as measured by the Vineland
Exploratory outcomes | Over 12 months post-infusion
  Change in quality of life, as measured by the Paediatric Quality of Life inventory
Exploratory outcomes | At 12 months post-infusion
  Quantification of viral vector integration in hepatocytes, from liver samples
Exploratory outcomes | Over 12 months post-infusion
  • Assessment of OTC enzymatic activity
Exploratory outcomes | Over 12 months post-infusion
  Assessment of vector genome copy numbers in liver samples

CONTACTS AND LOCATIONS:
Overall Officials: Federicco Mingozzi, Study Chair — Genethon
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Written requests will be considered by the HORACE Trial Management Group.